CLINICAL TRIAL: NCT00901381
Title: Open Prospective Randomized Controlled Trial of Efficacy and Safety of Granulocyte-colony Stimulating Factor Leukostim for Acute Ischemic Stroke.
Brief Title: Granulocyte-colony Stimulating Factor for Stem Cells Therapy for Acute Ischemic Stroke
Acronym: STEMTHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Institute of the Brain, Russia (Other)
Collaborators: Institute of Medical Cells Technologies (Unknown); City Hospital No 40, Saint Petersburg, Russia (Other)
Responsible Party: Andrey Belkin, Clinical Institute of the Brain, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GKSF-8
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Stem cells; Colony-stimulating factors; Filgrastim; Randomized controlled trial
MeSH Terms: conditions — Ischemic Stroke | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (Experimental)
  Interventions: Drug: Filgrastim
- Control (No Intervention)

INTERVENTIONS:
Drug: Filgrastim — 10 µg/kg subcutaneously once daily x 5 days
  Other Names: Leukostim
  Arms: G-CSF

SUMMARY:
The aim of the study is to investigate treatment with Leukostim (Filgrastim; granulocyte-colony stimulating factor; G-CSF) for acute ischemic stroke.

DETAILED DESCRIPTION:
Stroke is one of the main reasons of mortality and morbidity all over the world. In economically developed countries stroke takes 2 or 3 place in the structure of morbidity and mortality. In animal models, it was shown that autological stem cells transplantation significantly increased perfusion of ischemic area and improved lost motor and sensor functions. Granulocyte-colony stimulating factor (G-CSF) was used in some clinical trials without following autological transplantation. However, there are no enough evidence-based proved results of G-GSF safety and effectiveness in acute ischemic stroke. In order to determine safety and efficiency of G-CSF administration together with conventional treatment and conventional intensive care protocol during acute ischemic stroke we organized this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 to 70 years old
* CT/MRI confirmed ischemic stroke in carotid area during 48 hours after the onset of clinical signs
* Level of conscious lower than 15 and higher than 8 points by the Glasgow Coma Scale
* Acute extremity paresis lower than 4 points by Medical Research Consul scale

Exclusion Criteria:

* Premorbid dependency (modified Rankin Scale > 0)
* Intracerebral hemorrhage
* Transitory ischemic attack
* Patients with previous stroke
* Any disorders, that can affect interpretation of results (e.g. psychiatric or movement disorders)
* Hematological diseases
* Coagulopathy
* Malignancy
* Pregnancy and lactation
* Organ dysfunction that would preclude tests required for this study
* Known allergic reaction to G-CSF or a component of G-CSF
* Patients that have received a cytokine within the last 1 month or are currently receiving a cytokine treatment

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Dependence assessed by the modified Rankin scale | 180 day

SECONDARY OUTCOMES:
Impairment assessed by the Medical Research Consul scale and National Institutes of Health Stroke Scale | 180 day
Disability assessed by the Barthel Index and Glasgow Outcome Scale | 180 day
Infarct size assessed by the magneto-resonance imaging | 180 day
Safety was assessed as mortality, incidence of hemorrhagic transformation and serious adverse events | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Andrey A Belkin, MD, PhD., Principal Investigator — Clinical Institute of the Brain, Russia
Locations (1):
- Clinical Institute of the Brain, Yekaterinburg, Russia

REFERENCES:
- See also: Publication with study results — http://www.ncbi.nlm.nih.gov/pubmed/24323654